CLINICAL TRIAL: NCT07085247
Title: The Role of Cutibacterium Acnes in the Development of Degenerative Lumbar Intervertebral Disc Disease and the Clinical Effect of Microdiscectomy
Brief Title: The Role of Cutibacterium Acnes in the Development of Degenerative Lumbar Intervertebral Disc Disease
Status: Recruiting | Type: Observational
Sponsor: Masaryk University (Other)
Collaborators: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: NW25J-10-00060
Record Dates: First submitted 2025-04-29; First posted 2025-07-25 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: Lumbar Disc Herniation; Lumbar Disc Degeneration; Cutibacterium Acnes; Low Back Pain
Keywords: Cutibacterium acnes; Degenerative disc disease; Low back pain; Microdiscectomy; Clinical outcome
MeSH Terms: conditions — Intervertebral Disc Displacement; Intervertebral Disc Degeneration; Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prospective: 1. Patient enrollment:
     We plan to prospectively enroll at least 400 patients with lumbar disc herniation indicated for lumbar microdiscectomy
  2. Preoperative data collection:
     Baseline epidemiological, radiological and clinical data including survey questionnaires will be collected from each patient.
  3. Peri-operative tissue collection:
     Peri-operatively collected tissue samples of the herniated intervertebral disc will be immediately sent for histological examination.
  4. Microbiological examination:
     The presence, quantification, phylotyping of C.acnes and other bacteria, including virulence factors and antimicrobial susceptibility in the collected disc tissue will be examined by a microbiologist.
  5. Post-operative follow-up visits:
  Post-operative clinical status will be assessed using questionnaires at follow-up visits at 6 weeks, 6, and 12 months after surgery
- retrospective: All patients in retrospective cohort have completed epidemiologic, MRI or CT, microbiological, and clinical data. The epidemiological data include age, gender, disc herniation relapse, epidural steroid injection before the surgery, body mass index (BMI), the lumbar segment of herniation, type of herniation, and physical workload. The clinical data include microbiological findings from perioperatively collected disc tissue, preoperative spinal MRI, preoperative and postoperative pain intensity according to the visual analog scale (VAS), and functional disability for low back pain quantified by the Oswestry Disability Questionnaire (ODQ). In this part of the project, microbiological findings will be studied together with radiological changes in preoperative MRI and clinical status before and after surgery.

SUMMARY:
The goal of this study is to clarify the role of the bacterium Cutibacterium acnes in the development of degenerative disc disease in patients with lumbar disc herniation who underwent microdiscectomy as part of their regular medical care.

DETAILED DESCRIPTION:
The project is divided into retrospective and prospective parts. The retrospective part will consist of data processing and analysis using our large cohort of patients enrolled during the previous studies. The prospective part will include a) patient enrollment, b) preoperative data collection, c) perioperative tissue collection, d) microbiological examination, e) postoperative follow-up visits, and f) data management and statistical analyses.

Retrospective data processing and analysis For the retrospective part of the project, the investigators plan to use the C. acnes database stored at the Department of Neurosurgery, St. Anne's University Hospital, Brno, Czech Republic. This database contains 1200 anonymized adult patients with symptomatic lumbar disc herniation scheduled for microdiscectomy between 2015 and 2024. These patients were enrolled during the research project entitled "Presence of the low-virulence bacterium Propionibacterium acnes in the intervertebral disc tissue as a cause of chronic back pain". Each patient signed informed consent forms before enrolling in this study, enabling future data analyses. According to our preliminary review, at least 400 patients of the retrospective cohort have completed epidemiologic, MRI, microbiological, and clinical data. The epidemiological data include age, gender, disc herniation relapse, epidural steroid injection before the surgery, body mass index (BMI), the lumbar segment of herniation, type of herniation, and physical workload. The clinical data include microbiological findings from perioperatively collected disc tissue, preoperative spinal MRI, preoperative and postoperative pain intensity according to the visual analog scale (VAS), and functional disability for low back pain quantified by the Oswestry Disability Questionnaire (ODQ). Although the data is available, no hypotheses between C. acnes positivity and clinical outcomes have yet been tested on the dataset. Therefore, in this part of the project, microbiological findings will be studied together with radiological changes in preoperative MRI and clinical status before and after surgery.

Prospective data cohort

Patient enrollment - the investigators plan to enrol at least 400 patients with lumbar disc herniation indicated for microdiscectomy at the Department of Neurosurgery, Faculty of Medicine, Masaryk University and St. Anne's University Hospital, Brno, Czech Republic. Patients indicated for lumbar microdiscectomy will be prospectively screened, and those who pass the inclusion and exclusion criteria will be asked to sign the Informed Consent form to be enrolled in the study.

Preoperative data collection - baseline epidemiological and clinical data such as age, gender, disc herniation relapse, epidural steroid injection before the surgery, body mass index (BMI), the lumbar segment of herniation, type of herniation, and physical workload will be collected from each patient. Degenerative changes in the intervertebral discs and adjacent spinal structures will be evaluated on MRI as part of a standard preoperative examination. Clinical data will be obtained during the preoperative clinical exam and from patients in the form of questionnaires, including a numerical scale for leg and back pain, the Oswestry questionnaire evaluating the impact of low back pain on activities of daily living, and the Short Form quality of life questionnaire - 36 (SF- 36) to examine the quality of life before surgery.

Perioperative tissue collection - all operations for herniated intervertebral discs in patients included in the project will be performed at the Department of Neurosurgery, Faculty of Medicine, Masaryk University, and St. Anne's University Hospital, Brno, Czech Republic. The surgical site will undergo a comprehensive preparation, including three meticulous applications of povidone-iodine or an adequate antiseptic in case of iodine allergy. The site will then be draped using a standard sterile technique. Common prophylactic antibiotics will be given preoperatively in a single intravenous dose in all cases, with the usual prophylactic antibiotic being cefazolin; clindamycin or vancomycin will be administered in case of allergy. The exact location of the skin incision will be guided by intraoperative fluoroscopy. In all cases, a posterior midline approach will be used. The Caspar-type self-retaining retractor will be placed, and the ligamentum flavum will be removed under an operating microscope using Penfield dissectors and Kerrison rongeurs. The nerve root and dural sac will be gently retracted, and the posterior longitudinal ligament will be incised at the site of the herniated disc. The disc herniation will be exposed and removed with the remnant fragments of the nucleus pulposus in the intervertebral space. To minimize contamination of tissue samples, they will be retained in a sterile sample cup, labeled, and transported to the Department of Microbiology at St. Anne's University Hospital, Brno, Czech Republic. Tissue samples ranging from 3x3x5 mm to 10x5x5 mm will be utilized immediately for microbiological processing.

Microbiological examination - based on the preliminary study, the investigators plan to process the samples (semi)quantitatively. The samples will be homogenized by disintegration in a stomacher. Subsequently, the samples will be inoculated onto suitable culture media and cultured aerobically and anaerobically with subsequent semi-quantitative evaluation of the results. The quantity of bacteria in the sample will be expressed as colony-forming units (CFU) in 1 g of the sample. C. acnes burden in the sample exceeding 103 CFU/gram (≥103 CFU/gram) will be considered a clinically significant finding; C. acnes burden below <102 CFU/gram will indicate contamination; ≥102 - <103 CFU/gram will be interpreted as a borderline result.

Taxonomic identification of isolated strains will be performed by matrix-assisted laser desorption/ionization time-of-flight mass spectrometry (MALDI-TOF MS) as well as conventional phenotypic methods (biochemical tests, microscopy, etc.). For the phylotyping of our isolates, the investigators will use the multiplex PCR. To assess the ability to form a biofilm, the investigators will use the microtiter plate-based assay. The assay needs to be optimized, particularly with regard to suitable culture conditions and suitable treatment of the adhesion surfaces (peptide coating). A CAMP factor will be tested using the CAMP test with Staphylococcus aureus (CCM 6188). Hemolytic activity will be assessed using the blood agar with washed sheep erythrocytes. The production of some other virulence factors, e.g., hyaluronidase decapsulation test, chondroitin sulfatase, hyaluronidase, deoxyribonuclease, gelatinase, phosphatase, and lecithinase, will also be monitored. Antimicrobial susceptibility testing will be performed using phenotypic methods, broth microdilution, and/or standardized disk diffusion methods, according to the European Committee on Antimicrobial Susceptibility Testing - EUCAST Antimicrobial Susceptibility Testing (available at https://www.eucast.org/ast_of_bacteria).

Postoperative follow-up visits - postoperative clinical condition and the overall outcome will be evaluated by patients using the same standardized exams and questionnaires as before the surgery (numerical pain scale for leg and back, the Oswestry questionnaire, the Short Form quality of life questionnaire - 36 (SF-36). In addition to the mentioned questionnaires, patients will evaluate the success of the surgical treatment using the modified MacNab criteria and their satisfaction with the surgical treatment using the North American Spine Society (NASS) patient satisfaction index. Follow-up on-site visits will be carried out according to the standards of the Department of Neurosurgery, Faculty of Medicine, Masaryk University and St. Anne's University Hospital, Brno, Czech Republic, 6 weeks (± 1week), 6 months (± 2weeks), and 12 months (± 2weeks) after the operation.

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 18 years
* MRI of the lumbosacral spine performed one month ± 2weeks before surgery showing a disc protrusion, herniation, or free nucleus pulposus sequestration
* matching physical examination findings including positive straight leg raise test, dermatomal sensory deficits, myotome motor deficits, and diminished deep tendon reflexes.

Exclusion Criteria:

* antibiotics or corticosteroid use the month before surgery
* ongoing bacterial or viral infection
* immunocompromised patient
* trauma
* undefined radiological mass
* inflammatory arthritis
* other rheumatologic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to enroll at least 400 patients with lumbar disc herniation indicated for microdiscectomy at the Department of Neurosurgery, Faculty of Medicine, Masaryk University and St. Anne's University Hospital, Brno, Czech Republic. Patients indicated for lumbar microdiscectomy will be prospectively screened, and those who pass the inclusion and exclusion criteria will be asked to sign the Informed Consent form to be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The effect of C. acnes on functional disability in patients after microdiscectomy. | 6 weeks (± 1week) after the operation.
  The primary aim is a questionnaire-based comparison of the dynamics of the functional limitations according to ODI score between patients with different C. acnes bacterial load and C. acnes isolates in the disc tissue following microdiscectomy.

SECONDARY OUTCOMES:
The effect of C. acnes on functional disability in patients after microdiscectomy. | 6 months (± 2weeks) after surgery.
  The primary aim is a questionnaire-based comparison of the dynamics of the functional limitations according to ODI score between patients with different C. acnes bacterial load and C. acnes isolates in the disc tissue following microdiscectomy.
The effect of C. acnes on functional disability in patients after microdiscectomy. | 12 months (± 2weeks) after the operation.
  The primary aim is a questionnaire-based comparison of the dynamics of the functional limitations according to ODI score between patients with different C. acnes bacterial load and C. acnes isolates in the disc tissue following microdiscectomy.
The effect of C. acnes on radicular pain in patients after microdiscectomy. | 6 weeks (± 1week) after the operation.
  The secondary aim is a questionnaire-based comparison of the dynamics of radicular pain according to NRS between groups with different C. acnes bacterial load and C. acnes isolates in the disc tissue c
The effect of C. acnes on radicular pain in patients after microdiscectomy. | 6 months (± 2weeks) after the operation.
  The secondary aim is a questionnaire-based comparison of the dynamics of radicular pain according to NRS between groups with different C. acnes bacterial load and C. acnes isolates in the disc tissue c
The effect of C. acnes on radicular pain in patients after microdiscectomy. | 12 months (± 2weeks) after the operation.
  The secondary aim is a questionnaire-based comparison of the dynamics of radicular pain according to NRS between groups with different C. acnes bacterial load and C. acnes isolates in the disc tissue c
The effect of C. acnes on low back pain in patients after microdiscectomy. | 6 weeks (± 1week) after the operation.
  The primary endpoint is a questionnaire-based comparison of the dynamics of low back pain according to NRS in patients with different C. acnes bacterial load and C. acnes isolates in the disc tissue following microdiscectomy.
The effect of C. acnes on low back pain in patients after microdiscectomy. | 6 months (± 2weeks) after the operation.
  The primary endpoint is a questionnaire-based comparison of the dynamics of low back pain according to NRS in patients with different C. acnes bacterial load and C. acnes isolates in the disc tissue following microdiscectomy.
The effect of C. acnes on low back pain in patients after microdiscectomy. | 12 months (± 2weeks) after the operation.
  The primary endpoint is a questionnaire-based comparison of the dynamics of low back pain according to NRS in patients with different C. acnes bacterial load and C. acnes isolates in the disc tissue following microdiscectomy.
The effect of C. acnes on quality of life in patients after microdiscectomy. | 6 weeks (± 1week) after the operation.
  The secondary aim is to compare the dynamics of overall health status using SF-36 questionnaire in patients after microdiscectomy with different C. acnes bacterial load and C. acnes isolates in the disc tissue.
The effect of C. acnes on quality of life in patients after microdiscectomy. | 6 months (± 2weeks) after the operation.
  The secondary aim is to compare the dynamics of overall health status using SF-36 questionnaire in patients after microdiscectomy with different C. acnes bacterial load and C. acnes isolates in the disc tissue.
The effect of C. acnes on quality of life in patients after microdiscectomy. | 12 months (± 2weeks) after the operation.
  The secondary aim is to compare the dynamics of overall health status using SF-36 questionnaire in patients after microdiscectomy with different C. acnes bacterial load and C. acnes isolates in the disc tissue.
The influence of C. acnes on the success of surgical treatment in patients after microdiscectomy. | 6 weeks (± 1week) after the operation.
  The secondary aim is a questionnaire-based comparison of success of surgical treatment according to MacNab criteria, between groups with different C. acnes bacterial load and C. acnes isolates in the disc tissue at different time intervals following microdiscectomy.
The influence of C. acnes on the success of surgical treatment in patients after microdiscectomy. | 6 months (± 2weeks) after the operation.
  The secondary aim is a questionnaire-based comparison of success of surgical treatment according to MacNab criteria, between groups with different C. acnes bacterial load and C. acnes isolates in the disc tissue at different time intervals following microdiscectomy.
The influence of C. acnes on the success of surgical treatment in patients after microdiscectomy. | 12 months (± 2weeks) after the operation.
  The secondary aim is a questionnaire-based comparison of success of surgical treatment according to MacNab criteria, between groups with different C. acnes bacterial load and C. acnes isolates in the disc tissue at different time intervals following microdiscectomy.
The influence of C. acnes on patient satisfaction after microdiscectomy. | 6 weeks (± 1week) after the operation.
  The secondary objective is to compare patient satisfaction with surgical treatment according to the NASS patient satisfaction index criteria, between groups with different C. acnes bacterial load and C. acnes isolates in disc tissue at different time intervals after microdiscectomy.
The influence of C. acnes on patient satisfaction after microdiscectomy. | 6 months (± 2weeks) after the operation.
  The secondary objective is to compare patient satisfaction with surgical treatment according to the NASS patient satisfaction index criteria, between groups with different C. acnes bacterial load and C. acnes isolates in disc tissue at different time intervals after microdiscectomy.
The influence of C. acnes on patient satisfaction after microdiscectomy. | 12 months (± 2weeks) after the operation.
  The secondary objective is to compare patient satisfaction with surgical treatment according to the NASS patient satisfaction index criteria, between groups with different C. acnes bacterial load and C. acnes isolates in disc tissue at different time intervals after microdiscectomy.
Presence of other bacteria in disc tissue and their effect on radicular pain in patients after microdiscectomy. | 6 weeks (± 1week) after the operation.
  Evaluation of the presence of other bacteria in disc tissue and their clinical significance using a questionnaire-based comparison of radicular pain according to NRS at different time intervals after microdiscectomy.
Presence of other bacteria in disc tissue and their effect on radicular pain in patients after microdiscectomy. | 6 months (± 2weeks) after the operation.
  Evaluation of the presence of other bacteria in disc tissue and their clinical significance using a questionnaire-based comparison of radicular pain according to NRS at different time intervals after microdiscectomy.
Presence of other bacteria in disc tissue and their effect on radicular pain in patients after microdiscectomy | 12 months (± 2weeks) after the operation.
  Evaluation of the presence of other bacteria in disc tissue and their clinical significance using a questionnaire-based comparison of radicular pain according to NRS at different time intervals after microdiscectomy
Presence of other bacteria in disc tissue and their effect on low back pain in patients after microdiscectomy | 6 weeks (± 1week) after the operation.
  Evaluation of the presence of other bacteria in disc tissue and their clinical significance using a questionnaire-based comparison of low back pain according to NRS at different time intervals after microdiscectomy.
Presence of other bacteria in disc tissue and their effect on low back pain in patients after microdiscectomy. | 6 months (± 2weeks) after the operation.
  Evaluation of the presence of other bacteria in disc tissue and their clinical significance using a questionnaire-based comparison of low back pain according to NRS at different time intervals after microdiscectomy.
Presence of other bacteria in disc tissue and their effect on low back pain in patients after microdiscectomy | 12 months (± 2weeks) after the operation.
  Evaluation of the presence of other bacteria in disc tissue and their clinical significance using a questionnaire-based comparison of low back pain according to NRS at different time intervals after microdiscectomy.
Presence of other bacteria in disc tissue and their effect on functional disability in patients after microdiscectomy. | 6 weeks (± 1week) after the operation.
  Evaluation of the presence of other bacteria in disc tissue and their clinical significance using a questionnaire-based comparison of functional disability according to ODI score at different time intervals after microdiscectomy.
Presence of other bacteria in disc tissue and their effect on functional disability in patients after microdiscectomy | 6 months (± 2weeks) after the operation.
  Evaluation of the presence of other bacteria in disc tissue and their clinical significance using a questionnaire-based comparison of functional disability according to ODI score at different time intervals after microdiscectomy.
Presence of other bacteria in disc tissue and their effect on functional disability in patients after microdiscectomy | 12 months (± 2weeks) after the operation.
  Evaluation of the presence of other bacteria in disc tissue and their clinical significance using a questionnaire-based comparison of functional disability according to ODI score at different time intervals after microdiscectomy.
Presence of other bacteria in disc tissue and their effect on the quality of life in patients after microdiscectomy. | 6 weeks (± 1week) after the operation.
  Evaluation of the presence of other bacteria in the disc tissue and their role in the success of surgical treatment using SF-36 questionnaire-based comparison at different time intervals after microdiscectomy.
Presence of other bacteria in disc tissue and their effect on the quality of life in patients after microdiscectomy. | 6 months (± 2weeks) after the operation.
  Evaluation of the presence of other bacteria in the disc tissue and their role in the success of surgical treatment using SF-36 questionnaire-based comparison at different time intervals after microdiscectomy.
Presence of other bacteria in disc tissue and their effect on the quality of life in patients after microdiscectomy. | 12 months (± 2weeks) after the operation.
  Evaluation of the presence of other bacteria in the disc tissue and their role in the success of surgical treatment using SF-36 questionnaire-based comparison at different time intervals after microdiscectomy.
Presence of other bacteria in disc tissue and their role in the success of surgical treatment in patients after microdiscectomy | 6 weeks (± 1week) after the operation.
  Evaluation of the presence of other bacteria in the disc tissue and their role in the success of surgical treatment using MacNab criteria at different time intervals after microdiscectomy.
Presence of other bacteria in disc tissue and their role in the success of surgical treatment in patients after microdiscectomy | 6 months (± 2weeks) after the operation.
  Evaluation of the presence of other bacteria in the disc tissue and their role in the success of surgical treatment using MacNab criteria at different time intervals after microdiscectomy.
Presence of other bacteria in disc tissue and their role in the success of surgical treatment in patients after microdiscectomy | 12 months (± 2weeks) after the operation.
  Evaluation of the presence of other bacteria in the disc tissue and their role in the success of surgical treatment using MacNab criteria at different time intervals after microdiscectomy.
The presence of other bacteria in disc tissue and their role in patient satisfaction after microdiscectomy | 6 weeks (± 1week) after the operation.
  Evaluation of the presence of other bacteria in disc tissue and their role in patient satisfaction with surgical treatment using the NASS patient satisfaction index at different time intervals following microdiscectomy.
The presence of other bacteria in disc tissue and their role in patient satisfaction after microdiscectomy | 6 months (± 2weeks) after the operation.
  Evaluation of the presence of other bacteria in disc tissue and their role in patient satisfaction with surgical treatment using the NASS patient satisfaction index at different time intervals following microdiscectomy.
The presence of other bacteria in disc tissue and their role in patient satisfaction after microdiscectomy | 12 months (± 2weeks) after the operation.
  Evaluation of the presence of other bacteria in disc tissue and their role in patient satisfaction with surgical treatment using the NASS patient satisfaction index at different time intervals following microdiscectomy.
Retrospective evaluation of the influence of different C. acnes bacterial load in disc tissue on preoperative radicular pain. | Processing of retrospective data up to one year after the start of the study.
  A retrospective evaluation of our cohort of more than a thousand patients enrolled in a prospective study evaluating the presence of C. acnes in intervertebral disc tissue collected during microdiscectomy. Comparison of patients with different bacterial loads of C. acnes in disc tissue and their effect on preoperative radicular pain according to NRS.
Retrospective evaluation of the effect of different C. acnes bacterial load in disc tissue on preoperative low back pain. | Processing of retrospective data up to one year after the start of the study.
  A retrospective evaluation of our cohort of more than a thousand patients enrolled in a prospective study evaluating the presence of C. acnes in intervertebral disc tissue collected during microdiscectomy. Comparison of patients with different bacterial loads of C. acnes in disc tissue and their effect on preoperative low back pain according to NRS.
Retrospective evaluation of the influence of different C. acnes bacterial load in disc tissue on preoperative functional disability | Processing of retrospective data up to one year after the start of the study
  A retrospective evaluation of our cohort of more than a thousand patients enrolled in a prospective study evaluating the presence of C. acnes in intervertebral disc tissue collected during microdiscectomy. Comparison of patients with different bacterial loads of C. acnes in disc tissue and their effect on preoperative functional disability according to ODI score.
Retrospective evaluation of the influence of different C. acnes bacterial load in disc tissue on the occurrence of Modic changes on preoperative MRI | Processing of retrospective data up to one year after the start of the study.
  A retrospective evaluation of our cohort of more than a thousand patients enrolled in a prospective study evaluating the presence of C. acnes in intervertebral disc tissue collected during microdiscectomy. Comparison of patients with different bacterial loads of C. acnes in disc tissue and their possible relationship with the occurrence of Modic changes on preoperative MRI.
Retrospective evaluation of the influence of different C. acnes bacterial load in disc tissue on the severity of degenerative changes in the intervertebral disc. | Processing of retrospective data up to one year after the start of the study
  A retrospective evaluation of our cohort of more than a thousand patients enrolled in a prospective study evaluating the presence of C. acnes in intervertebral disc tissue collected during microdiscectomy. Comparison of patients with different bacterial loads of C. acnes in disc tissue and their possible relationship with the severity of intervertebral disc degeneration according to Pfirrmann score.
Retrospective evaluation of the influence of different C. acnes bacterial load in disc tissue on the severity of vertebral endplate damage. | Processing of retrospective data up to one year after the start of the study.
  A retrospective evaluation of our cohort of more than a thousand patients enrolled in a prospective study evaluating the presence of C. acnes in intervertebral disc tissue collected during microdiscectomy. Comparison of patients with different bacterial loads of C. acnes in disc tissue and their possible relationship with the severity of vertebral endplate damage according to Endplate Damage Score.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Anne´s University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No